CLINICAL TRIAL: NCT01347944
Title: Observational, Non-interventional, Multicenter Study Aimed at Collecting Retrospective/Prospective 648/96 Italian Registry Data Related to Lenalidomide (Revlimid®) Prescription to Patients With Myelodysplastic Syndromes
Brief Title: MORE - Monitoring Revlimid - Collecting of Patient Information From Myelodysplastic Syndrome (MDS) Italian National Registry
Acronym: MORE
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIPMS- Celgene-MDS-ITA-002
Record Dates: First submitted 2010-10-29; First posted 2011-05-05 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndrome
Keywords: MORE; Monitoring Revlimid; Myelodysplastic Syndrome; Transfusion-dependent anemia; 5q deletion; lenalidomide
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: lenalidomide — Patients who were prescribed Revlimid from 31October 2008 to present.
  Other Names: Revlimid®

SUMMARY:
The purpose of this study is to collect clinical and laboratory data for patients affected by intermediate 1 and low risk Myelodysplastic Syndrome (MDS) associated by deletion 5q who were prescribed Revlimid from 31October 2008 to present. Revlimid is available in Italy for these patients since October 2008 based on a local disposition of the Italian Drug Agency (AIFA) issued according to a National law named 648/96.

DETAILED DESCRIPTION:
There will be retrospective collection and integration of clinical laboratory data as well as prospective data collection on the same patients.

ELIGIBILITY:
Inclusion Criteria:

* intermediate 1 and low risk MDS patients associated with:

  1. transfusion dependency anemia (at least 2 units per 8 weeks before starting of Revlimid treatment )
  2. 5q31-33 deletion isolated or associated to other chromosomal abnormalities.

     Exclusion Criteria:
* patients with serum creatinine > 2.5mg/dl
* child bearing potential females who do not use adequate contraceptive methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by intermediate-1 and low risk MDS associated by deletion 5q who were prescribed Revlimid from 31October 2008 to present.
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects achieving red blood cell (RBC) transfusion independence | 14 months
Number of subjects achieving an erythroid response | 14 months
Number of subjects achieving a cytogenetic response | 14 months

SECONDARY OUTCOMES:
Number of participants with adverse events | 14 months
Duration of RBC transfusion independence | 14 months
Duration of cytogenetic response | 14 months
Time to RBC transfusion independence | 14 months
Progression to acute myeloid leukemia (AML) | 14 months
Number of participants alive | 14 months

CONTACTS AND LOCATIONS:
Overall Officials: Sante Cundari, PhD, MSc, Study Director — Celgene s.r.l.
Locations (45):
- Italy (45):
  - Dipartimento Onco - Ematologico Azienda Ospedaliera SS Antonio, Biagio e Cesare Arrigo, Alessandria
  - Unità Operativa Clinica di Ematologia Azianda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Dipartimento di Oncologia Medica Ospedale Cardinale G. Massaia, Asti
  - Ematologia Azienda Ospedaliera Universitaria Policlinico di Bari, Bari
  - Dipartimento di Ematologia Ospedale dell'U.L.S.S. n.1 Belluno, Belluno
  - Ematologia A.O. Ospedale Riuniti di Bergamo, Bergamo
  - Dip. Medicina Interna Ospedale degli Infermi di Biella, Biella
  - Dipartimento di Ematologia Spedale Civili di Brescia, Brescia
  - Dipartimento Trapianto di Midollo Allogenico Spedale Civili di Brescia, Brescia
  - Dipartimento di Ematologia Ospedale R. Binaghi, Cagliari
  - Dip. Di Oncoematologia A.O. S.Anna e S. Sebastiano, Caserta
  - Dip. Di Ematologia A.O. Istituti Ospedalieri, Cremona
  - Dip. Di Ematologia Az. Ospedaliero-Universitaria Careggi, Florence
  - Dip. Di Ematologia A.O. Universitaria S. Martino, Genova
  - Dip. Di Medicina Interna A.O. Universitaria S. Martino, Genova
  - Dip. Di Ematologia Azienda Ospedaliera V. Fazzi, Lecce
  - Centro Trapianti di Midollo Ospedale Maggiore Policlinico, Milan
  - Dip. Di Ematologia Policlinico, Az. Ospedaliero- Universitaria, Modena
  - Dip. Di Ematologia Azienda Ospedaliera S. Gerardo, Monza
  - Dip. Di Oncoematologia A.O. Universitaria Federico II, Napoli
  - Dip. Di Ematologia Presidio Ospedaliero Umberto I, Nocera Inferiore
  - Dip. Di Ematologia Ospedale S. Francesco, Nuoro
  - Dip. Di Ematologia Azienda Ospedaliera, Padua
  - Dip. di Ematologia Azienda Ospedaliera, Parma
  - Dip. Di Ematologia Azienda Ospedaliera - Osp. S. Maria della Misericordia, Perugia
  - Dip. Di Ematologia Azienda Ospedaliera s. Salvatore, Pesaro
  - Dip. Di Ematologia Az. Ospedaliera Regionale S. Carlo, Potenza
  - Servizio di Ematologia - Dip. di Oncologia Az. Ospedaliera di Reggio Emilia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Dip. Di Ematologia Ospedale S. Maria delle Croci, Revenna
  - U. O. Ematologia Az. Ospedaliero-Universitaria Policlinico Tor Vergata, Roma
  - U.O.C Ematologia Ospedale S. Eugenio, Piazzale dell'Umanesimo, Roma
  - Dip. di Ematologia Policlinico Umberto I, Roma
  - U.O.C. Ematologia Policlinico Universitario Gemelli, Roma
  - Dip. di Oncoematologia Ospedale Civile Giannettasio, Rossano
  - Dip. di Oncoematologia Az. ULSS 18, Rovigo
  - Struttura di Ematologia, Dip. di Oncoematologia IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Dip. di Ematologia Policlinico Universitario di Sassari, Sassari
  - Divisione di Ematologia e Trapianti Spedali Riuniti, Siena
  - Dip. di Ematologia 1 A.O. Universitaria S.Giovanni Battista, Torino
  - Dip. di Ematologia 2 A.O. Universitaria S.Giovanni Battista, Torino
  - Dip. di Ematologia e Terapie Cellulari Ospedale Mauriziano Umberto I, Torino
  - Unità Operativa Trasfusionale ed Immunologia Centro di riferimento per le malattie rare e centro regionale per le malattie del sangue Ospedale S. Giacomo Apostolo, Treviso
  - Ospedale Dell'Angelo USL12 - Venezia (Mestre), Venezia
  - Dip. Funzionale di Terapie Cellulari e Ematologia Azienda Sanitaria ULSS 6 - Osp. di Vicenza, Vicenza
  - Dip. Di Ematologia Ospedale di Belcolle, Viterbo

REFERENCES:
- [Background] Arcioni F, Roncadori A, Di Battista V, Tura S, Covezzoli A, Cundari S, Mecucci C; MORE Study Centres. Lenalidomide treatment of myelodysplastic syndromes with chromosome 5q deletion: Results from the National Registry of the Italian Drug Agency. Eur J Haematol. 2018 Jul;101(1):78-85. doi: 10.1111/ejh.13067. Epub 2018 May 22. PMID 29569278